CLINICAL TRIAL: NCT02964052
Title: Selection Criteria in Endovascular Thrombectomy and Thrombolytic Therapy (SECRET) Study: Development of Patient Selection Criteria Using CT Images and Accompanying Diseases for Efficient Intravenous Thrombolytic and Intra-arterial Recanalization Therapy in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-1196
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke patients: Acute ischemic stroke patients who received intravenous (IV) thrombolysis and/or intra-arterial (IA) recanalization treatment
  Interventions: Other: Brain CT imaging

INTERVENTIONS:
Other: Brain CT imaging — Investigators will analyzed the CT image that was performed in patients with hyperacute stroke. The CT protocol includes CT thrombus, collateral, core images. Investigators also obtain detailed history and laboratory and imaging result for comorbidity. The comorbidity index protocol is based on the Charlson comorbidity index.

SUMMARY:
Use of intravenous (IV) thrombolysis and intra-arterial (IA) recanalization treatment has been rapidly increasing, However, despite of the treatment, recanalization rates are 22.6 - 70% and only 30-50% of patients show meaningful clinical improvements. Mechanisms of futile recanalization may include 1) large ischemic core, 2) poor collateral, and 3) presence of comorbidity. In this regards, developing selection criteria using acute stroke imaging and comorbidity is warranted.

Investigators will recruit the consecutive acute stroke patients who received IV thrombolysis and/or IA recanalization treatment. This study will perform with prospective design to develop CT-based clot, core and collateral scores and a comorbidity index for selecting stroke patients who are at high risks by the treatment. Investigators will firstly establish the CT-based scores and comorbidity index using a pre-existing cohort database. Using these CT-based and comorbidity index, Investigators will validate them in a multi-center prospectively cohort. In addition, Investigators will assess the cost-effectiveness of selecting patients based on the comorbidity index.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old
* Acute ischemic stroke patients who underwent CT angiographies before IV thrombolysis and/or IA recanalization treatment
* Patients who give an informed consents for participation in the study or the legal representative or immediate family give informed consent on behalf of patients in case of difficulty to decide study enrollment.

Exclusion Criteria:

* Age <20 years old
* Acute ischemic stroke patients who did not receive IV thrombolysis and/or IA recanalization treatment
* No informed consents from patients

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients who received intravenous (IV) thrombolysis and/or intra-arterial (IA) recanalization treatment
Sampling Method: Probability Sample
Enrollment: 1359 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale scores | 3 months after discharge day
Death | 6 months after discharge day
National Institutes of Health Stroke Scale (NIHSS) scores | 1 hr after IV rt-PA infusion
Recanalization rate | after 16 hrs thrombolytic treatments in MRA, CTA, or digital subtraction angiography (DSA)
Recanalization rate | after 24 hrs thrombolytic treatments in MRA, CTA, or digital subtraction angiography (DSA)
Recanalization rate | after 32 hrs thrombolytic treatments in MRA, CTA, or digital subtraction angiography (DSA)
Symptomatic hemorrhagic transformation rate | after 16 hrs thrombolytic treatments in MR or CT
Symptomatic hemorrhagic transformation rate | after 24 hrs thrombolytic treatments in MR or CT
Symptomatic hemorrhagic transformation rate | after 32 hrs thrombolytic treatments in MR or CT
asymptomatic hemorrhagic transformation rate | after 16 hrs thrombolysis in MR or CT
asymptomatic hemorrhagic transformation rate | after 24 hrs thrombolysis in MR or CT
asymptomatic hemorrhagic transformation rate | after 32 hrs thrombolysis in MR or CT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam HS, Kim YD, Yoo J, Park H, Kim BM, Bang OY, Kim HC, Han E, Kim DJ, Lee IH, Lee H, Choi JK, Lee KY, Lee HS, Shin DH, Choi HY, Sohn SI, Hong JH, Lee JY, Baek JH, Kim GS, Seo WK, Chung JW, Kim SH, Song TJ, Han SW, Park JH, Kim J, Jung YH, Cho HJ, Ahn SH, Seo KD, Lee KO, Song J, Heo JH. d-Dimer Level After Endovascular Treatment Can Help Predict Outcome of Acute Ischemic Stroke. Stroke Vasc Interv Neurol. 2023 Feb 25;3(3):e000713. doi: 10.1161/SVIN.122.000713. eCollection 2023 May. PMID 41584989
- [Derived] Kim HJ, Park MS, Yoo J, Kim YD, Park H, Kim BM, Bang OY, Kim HC, Han E, Kim DJ, Heo J, Choi JK, Lee KY, Lee HS, Shin DH, Choi HY, Sohn SI, Hong JH, Lee JY, Baek JH, Kim GS, Seo WK, Chung JW, Kim SH, Han SW, Park JH, Kim J, Jung YH, Cho HJ, Ahn SH, Lee SI, Seo KD, Chang Y, Song TJ, Nam HS; SECRET Study Investigators. Association between CHADS2, CHA2DS2-VASc, ATRIA, and Essen Stroke Risk Scores and Unsuccessful Recanalization after Endovascular Thrombectomy in Acute Ischemic Stroke Patients. J Clin Med. 2022 Jan 5;11(1):274. doi: 10.3390/jcm11010274. PMID 35012015